CLINICAL TRIAL: NCT07177807
Title: Clinical Characteristics of Neovascular Glaucoma : A Six-Year Retrospective Study
Brief Title: Clinical Characteristics of Neovascular Glaucoma
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Collaborators: The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Central Hospital of Xiaogan (Other)
Responsible Party: Sponsor
Other Study IDs: 20250719
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Neovascular Glaucoma
Keywords: Neovascular glaucoma; clinical feature; Retinal Vein Occlusion; Diabetic Retinopathy
MeSH Terms: conditions — Glaucoma, Neovascular; Retinal Vein Occlusion; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALL group
- DR group
- RVO group

SUMMARY:
The goal of this observational study is to explore the clinical characteristics of patients with neovascular glaucoma (NVG), and to analyze the relationship between NVG and various underlying diseases, ocular conditions, lifestyle, inflammatory markers, and treatment response. To systematically analyze the clinical data of NVG patients with different types of primary disease, further reveal the different clinical characteristics of NVG patients with different primary disease, and describe the selection of treatment methods in recent years, in order to provide more scientific basis for clinical treatment.

DETAILED DESCRIPTION:
The goal of this observational study is to explore the clinical characteristics of patients with neovascular glaucoma (NVG), and to analyze the relationship between NVG and various underlying diseases, ocular conditions, lifestyle, inflammatory markers, and treatment response. To systematically analyze the clinical data of NVG patients with different types of primary disease, further reveal the different clinical characteristics of NVG patients with different primary disease, and describe the selection of treatment methods in recent years, in order to provide more scientific basis for clinical treatment.Patients discharged from multiple hospitals from January 2018 to September 2024 with the diagnosis of NVG were retrospectively investigated. The medical history of each patient was reviewed, and the basic information, past medical history, eye examinations and their results, treatment plans, and prognosis information of the patients were recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the diagnostic criteria for NVG.

Exclusion Criteria:

* Patients with incomplete clinical data and information.
* Severe systemic diseases (such as chronic renal failure requiring dialysis, severe neurological diseases, immune diseases), pregnancy or lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients with NVG diagnosed by ophthalmic examination in the Second Clinical Hospital of Wuhan University, Central Hospital of Enshi Tujia and Miao Autonomous Prefecturefrom and Central Hospital of Xiaogan from January 2018 to September 2024 were enrolled.
  A certain number of healthy volunteers in the Physical Examination Center of the Second Clinical Hospital of Wuhan University from January 2018 to September 2024 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | Time Frame: Pre-operative, post-operative follow-up at 1 month, 3 months, 6 months, 1 year, etc.
  best-corrected visual acuity （BCVA）
intraocular pressure | Time Frame: Pre-operative, post-operative follow-up at 1 month, 3 months, 6 months, 1 year, etc.
  intraocular pressure(IOP)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China